CLINICAL TRIAL: NCT07037862
Title: A 2-Part, Randomized, Double-Blind, Placebo-Controlled Study in Participants With Duchenne Muscular Dystrophy Amenable to Exon 44 Skipping With an Initial Multiple Ascending Dose Part A to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ENTR-601-44, Followed by Part B to Evaluate the Safety and Efficacy of ENTR-601-44 (ELEVATE-44)
Brief Title: A Study in Participants With Duchenne Muscular Dystrophy Amenable to Exon 44 Skipping to Evaluate the Safety and Efficacy of ENTR-601-44
Acronym: ELEVATE-44
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Entrada Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ENTR-601-44-201; 2024-517584-23-00 (EU CTIS Number); U1111-1316-5469 (Other: WHO)
Record Dates: First submitted 2025-05-01; First posted 2025-06-26 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
Keywords: Duchenne Muscular Dystrophy; DMD; exon skipping therapy; oligonucleotide therapy
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ENTR-601-44 (Experimental): intravenous infusion every 6 weeks
  Interventions: Drug: ENTR-601-44
- Placebo (Placebo Comparator): intravenous infusion every 6 weeks
  Interventions: Drug: ENTR-601-44 - matching placebo

INTERVENTIONS:
Drug: ENTR-601-44 — intravenous infusion
  Arms: ENTR-601-44
Drug: ENTR-601-44 - matching placebo — intravenous infusion
  Arms: Placebo

SUMMARY:
This is a study of the investigational medicine ENTR-601-44 in participants who have Duchenne muscular dystrophy (DMD), a rare genetic condition.

The researchers want to: Test how safe ENTR-601-44 is, learn about any side effects, and look at the potential positive effects of ENTR-601-44, compared to placebo. Placebo looks like the investigational medicine but does not contain any active ingredient. In this summary ENTR-601-44 and placebo are both called study treatments.

The study has 2 parts: Part A: to evaluate if ENTR-601-44 is safe and to determine the best dose of ENTR-601-44 for Part B. Part B: to further evaluate the effect and safety of ENTR-601-44 at the dose determined in Part A.

Participants will be able to roll into an open-label treatment period during which the safety and efficacy of extended dosing will be evaluated.

Participants will:

* Receive study treatment in the form of multiple intravenous (IV) infusions (slow injection) into a vein over the course of several weeks in Part A and in Part B
* Visit the clinic regularly for checkups and tests such as: blood and urine tests, physical examinations, questionnaires, and exercise tests. Participants will have a muscle biopsy at the beginning of their participation and after their last dose to allow researchers to compare whether there have been changes in the muscle as a result of the study drug.

Participants are allowed to continue receiving their standard of care therapy for DMD during the study, as long as their health remains stable.

ELIGIBILITY:
Principal inclusion criteria

1. Genetic diagnosis of Duchenne muscular dystrophy (DMD) and confirmed pathologic variant in the dystrophin gene amenable to exon 44 skipping as reviewed by a central genetic counselor.
2. Assigned male at birth with clinical signs compatible with Duchenne muscular dystrophy as determined by the investigator.
3. Part A: 4-20 years of age, inclusive.
4. Ambulatory Status Part A: ambulatory with a Performance of the Upper Limb v2.0 (PUL 2.0) Entry as per protocol at Screening
5. Adequate muscle for obtaining tissue biopsy as assessed by the investigator.
6. Other protocol-defined criteria apply.

Principal exclusion criteria

1. Any significant concomitant medical condition that might interfere with the ability to comply with protocol requirements.
2. Has an acute illness within 4 weeks prior to the first dose of study drug which may interfere with study measurements or jeopardize participant's safety.
3. Use of the following medications:

   1. Prior treatment with any exon skipping therapy at any time
   2. Prior treatment with any gene therapy at any time
   3. Use of anti-coagulants, anti-thrombotics, or anti-platelet agents
   4. Use of an immunosuppressants (other than oral corticosteroids for DMD conditions)
   5. Has taken or is currently taking a histone deacetylase (HDAC) inhibitor, including (but not limited to) givinostat
4. Laboratory abnormalities.
5. Daytime ventilator dependence or any use of invasive mechanical ventilation via tracheostomy.
6. Has an abnormal electrocardiogram (ECG) reading assessed as clinically significant by the investigator, and/or a QT interval with Fridericia correction method (QTcF) >450 msec at Screening or prior to the first dose of study drug on Day 1.
7. Received any experimental or investigational drug, etc. within 3 months prior to first dose or within 5 half-lives (whichever is longer).
8. Other protocol-defined criteria apply.

Ages: 4 Years to 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 24 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2029-03-28 (Estimated); Study Completion 2029-03-28 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Treatment Emergent Adverse Events (TEAEs) according to study protocol (Part A and Open Label (OL) Period) | From baseline through End of Study (up to 62 weeks).
  Safety will be assessed by monitoring adverse events, physical examination, vital signs and clinical laboratory tests.

SECONDARY OUTCOMES:
Plasma, muscle, and urine concentration of ENTR-601-44 and its final metabolite (Part A and Open Label (OL) Period) | From Baseline through End of Study (up to 62 weeks).
Change from baseline to End of Part A in dystrophin by Western blot from muscle biopsy (Part A) | Baseline, End of Part A (up to 25 weeks)
Change from baseline to End of Part A in dystrophin expression and localization from muscle biopsy (Part A) | Baseline, End of Part A (up to 25 weeks)
Percent change from baseline to End of Part A in exon 44 skipping measured in muscle biopsy at End of Study (Part A) | Baseline, End of Part A (up to 25 weeks)
Anti-drug antibody (ADA) and anti-dystrophin antibody in serum (Part A and OL Period) | From baseline through End of Study (up to 62 weeks).
Change from baseline to End of OL Period in 10-Meter Walk/Run (10MWR) (Part A and OL Period) | Baseline, End of Study (up to 62 weeks)
Change from baseline to End of OL Period in Timed Rise from Floor (Part A and OL Period) | Baseline, End of Study (up to 62 weeks)
Change from baseline to End of OL Period in Timed 4-Stair Climb (4SC) (Part A and OL Period) | Baseline, End of Study (up to 62 weeks).
Change from baseline to End of OL Period in 95th centile Stride Velocity (SV95C) (Part A and OL Period) | Baseline, End of Study (up to 62 weeks)
Change from baseline to End of OL Period in North Star Ambulatory Assessment (NSAA) (Part A and OL Period) | Baseline, End of Study (up to 62 weeks)
  Ordinal scale with 0 as the minimum score and 34 as the maximum score (higher score - better outcome).
Change from baseline to End of OL Period in Performance of the Upper Limb v2.0 (PUL 2.0) (Part A and OL Period) | Baseline, End of Study (up to 62 weeks)
  Ordinal scale with 0 as the minimum score and 42 as the maximum score (higher score - better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Entrada Therapeutics Clinical Trials, Study Director — Entrada Therapeutics, Inc.
Locations (15):
- Belgium (3):
  - University Hospital Gent, Ghent
  - UZ Leuven, Leuven
  - Centre Hospitalier Régional de la Citadelle, Liège
- Italy (4):
  - IRCCS Ospedale San Raffaele, Milan
  - Fondazione Serena Onlus - Centro Clinico NeMO Milano, Milan
  - Ospedale Pediatrico Bambino Gesu, Rome
  - Fondazione Policlinico Universitario A. Gemelli IRCCS - Universita Cattolica del Sacro Cuore, Rome
- Spain (2):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital Sant Joan de Deu, Barcelona
- United Kingdom (6):
  - Leeds General Infirmary, Leeds
  - Alder Hey Children's NHS Foundation Trust, Liverpool
  - Great Ormond Street Hospital for Children, London
  - Royal Manchester Children's Hospital, Manchester
  - Freeman Hospital, Newcastle upon Tyne
  - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: No
The datasets generated during and/or analysed during the current study are not expected to be made available due to due to the data's high commercial sensitivity.